CLINICAL TRIAL: NCT01933724
Title: The Assessment of Prednisone In Remission Trial (TAPIR) - Patient Centric Approach
Acronym: TAPIR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCRC 5526B TAPIR; 5526B (Other: VCRC); R01HL115041 (NIH)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Granulomatosis With Polyangiitis; Wegener Granulomatosis; Vasculitis
Keywords: granulomatosis with polyangiitis; GPA; Wegeners'; WG; vasculitis; taper; prednisone; glucocorticoid; ANCA-associated vasculitis; AAV; Wegener Granulomatosis; Systemic Vasculitis; Lung diseases, interstitial; Lung diseases; Respiratory Tract Diseases; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vascular Diseases; Cardiovascular Diseases; Glucocorticoids; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Pharmacologic Actions; Antineoplastic Agents, Hormonal; Antineoplastic Agents; Therapeutic Uses; Anti-Inflammatory Agents
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Systemic Vasculitis; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Prednisone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg prednisone (Experimental): Subjects will be randomized to 5 mg per day of prednisone for a 6 month period.
  Interventions: Drug: 5 mg prednisone
- 0 mg prednisone (Experimental): Subjects will be randomized to 0 mg per day of prednisone dose for a 6 month period.
  Interventions: Drug: 0 mg prednisone

INTERVENTIONS:
Drug: 5 mg prednisone — Subjects will be randomized to take 5 mg per day of prednisone for a 6 month period.
  Other Names: 5 mg glucocorticoids; 5 mg/day prednisone
  Arms: 5 mg prednisone
Drug: 0 mg prednisone — Subjects will be randomized to taper their prednisone dose to no prednisone for a 6 month period.
  Other Names: no prednisone; no glucocorticoids
  Arms: 0 mg prednisone

SUMMARY:
This is a randomized controlled trial in patients with a diagnosis of granulomatosis with polyangiitis (GPA; Wegener's)that are in remission to evaluate the effects of using low-dose glucocorticoids ( 5 mg/day of prednisone) as compared to stopping glucocorticoid treatment entirely (0 mg/day of prednisone)on rates of disease relapse/disease flares.

This study is a novel approach to conducting a randomized clinical trial in the community setting. This study is being conducted in parallel with a similar study at established vasculitis institutions. This study will have a patient centric approach to research in that subjects will be recruited online and through social media and vasculitis support networks. Participants will be consented online and will receive care through their regular treating physician so no travel or additional doctor visits are required. Study participants will consent to the study and complete online questionnaires about their prednisone dose and about how they are feeling.

DETAILED DESCRIPTION:
This open label pilot study will randomize 60 participants with GPA in remission affecting the sinonasal tract, oral mucosa, skin, musculoskeletal system, pulmonary parenchyma, or other disease features that warranted an administration of 20 mg/day or more within the last 12 months. At the time of enrollment, participants will need to be taking prednisone at a dose of ≥ 5mg/day and ≤ 20 mg/day. All enrolled participants will be instructed to reduce the daily dose of prednisone according to their treating physician. Once participants reach a prednisone dose of 5mg/day, they will be randomized at a 1:1 ratio to continue prednisone at 5 mg/day or to taper prednisone to 0 mg/day. Participants will be followed for approximately six months from reaching a prednisone dose of 5 mg/day.

The primary study outcome is the proportion of participants who increase prednisone for disease relapse within 6 months of randomization. Participant data collected via this study will be combined with that from a complementary study conducted at Vasculitis Clinical Research Consortium (VCRC) clinical centers.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of granulomatosis with polyangiitis (GPA) (verified by medical record review by the Protocol Oversight Management Team) where patients will need to meet at least 2 of the 5 for the classification of GPA, at least one of which must be criterion d or e.

   The modified American College of Rheumatology (ACR) criteria are:
   1. Nasal or oral inflammation, defined as the development of painful or painless oral ulcers or purulent or bloody nasal discharge
   2. Abnormal chest radiograph, defined as the presence of nodules, fixed infiltrates, or cavities.
   3. Active urinary sediment, defined as microscopic hematuria (>5 red blood cells per high power field) or red blood cell casts
   4. Granulomatosis inflammation on biopsy, defined as histologic changes showing granulomatous inflammation within the wall of an artery or in the perivascular or extravascular area. Note: Pauci-immune glomerulonephritis seen on kidney biopsy will suffice for this criterion.
   5. Positive anti-neutrophil cytoplasmic antibody (ANCA) test specific for proteinase-3 measures by enzyme-linked immunoassay Patients who are myeloperoxidase (MPO) positive or ANCA negative are still eligible for this study if they meet the criteria above and are felt to have GPA.
2. Active disease within the prior 12 months (initial presentation or relapse) that at time of active disease required treatment with prednisone ≥ 20 mg/day
3. Disease remission at time of enrollment
4. Prednisone dose at time of enrollment of ≥ 5mg/day and ≤ 20 mg/day
5. Participant age of 18 years or greater
6. If the patient is taking an immunosuppressive medication agent other than prednisone (maintenance agent) then the maintenance agent must be at a stable dose for one month prior to enrollment with no plans by the treating physician to change the dose (other than for safety purposes/toxicity) for the duration of the study (through the month 6 visit or early termination). Acceptable maintenance agents include azathioprine, leflunomide, 6-mercaptopurine, methotrexate, mycophenolate mofetil, rituximab, or mycophenolate sodium. Patients may be on trimethoprim/sulfamethoxazole (TMP/SMX) for use as either a maintenance agent or for prophylaxis for infection. TMP/SMX may be used in combination with other drugs.

   6.1 If the patient is regularly taking trimethoprim/sulfamethoxazole at any dose then the patient is eligible if there no plans by the treating physician to change the dose after enrollment (other than for dose reduction or discontinuation for safety purposes/toxicity) for the duration of the study.
7. Agreement from Treating Physician that 0mg/day of prednisone or 5mg/day of prednisone is standard of care
8. Participant's Treating Physician is located in the United States

Exclusion Criteria:

1. Comorbid condition that has moderate likelihood of requiring a course of prednisone within one year of enrollment (e.g. chronic obstructive pulmonary disease (COPD), asthma, adrenal insufficiency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prednisone dose increase for disease relapse | 6 months
  Physician decision to increase prednisone dose for GPA disease relapse

SECONDARY OUTCOMES:
Rates of disease flare sub types | 6 months
  Rates of GPA disease flare sub types: severe versus non-severe
Time to event flare | 6 months
  Time from randomization to GPA disease flare
Health related quality of life | 6 months
  Health related quality of life as assessed through the Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire
Safety Outcomes | 6 months
  Serious adverse events and infections
Protocol performance | 6 months
  * Patient characteristics
  * Protocol compliance This study is being conducted in parallel to a study at VCRC clinical centers. Protocol performance will be assessed through comparison of participant retention, data completeness, timeliness of data entry, and data accuracy between the two studies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Merkel, MD, MPH, Principal Investigator — University of Pennsylvania; Jeffrey P Krischer, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida TAPIR Study Team, Tampa, Florida, United States

REFERENCES:
- [Result] Krischer J, Cronholm PF, Burroughs C, McAlear CA, Borchin R, Easley E, Davis T, Kullman J, Carette S, Khalidi N, Koening C, Langford CA, Monach P, Moreland L, Pagnoux C, Specks U, Sreih AG, Ytterberg S, Merkel PA; Vasculitis Clinical Research Consortium. Experience With Direct-to-Patient Recruitment for Enrollment Into a Clinical Trial in a Rare Disease: A Web-Based Study. J Med Internet Res. 2017 Feb 28;19(2):e50. doi: 10.2196/jmir.6798. PMID 28246067
- [Derived] Cronholm PF, Applequist J, Krischer J, Fontenot E, Davis T, Burroughs C, McAlear CA, Borchin R, Kullman J, Carette S, Khalidi N, Koening C, Langford CA, Monach P, Moreland L, Pagnoux C, Specks U, Sreih AG, Ytterberg SR, Merkel PA; Vasculitis Clinical Research Consortium. A study of implementation factors for a novel approach to clinical trials: constructs for consideration in the coordination of direct-to-patient online-based medical research. BMC Med Res Methodol. 2024 Oct 18;24(1):244. doi: 10.1186/s12874-024-02352-w. PMID 39425055

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT01933724/Prot_SAP_000.pdf